CLINICAL TRIAL: NCT03863249
Title: Use of the xCELLigence System for Quantification of Bacterial Biofilm's Real Time Formation and Antibiotics Selection: Randomized Clinical Trial.
Brief Title: Use of the xCELLigence System for Quantification of Bacterial Biofilm's Real Time Formation and Antibiotics Selection.
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Valencia (Other)
Collaborators: Centro Superior de Investigación en Salud Publica (Other Government); Fundación para el Fomento de la Investigación Sanitaria y Biomédica de la Comunitat Valenciana (Other)
Responsible Party: Principal Investigator, Andres Lopez Roldan, Associate professor, University of Valencia
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: UV4
Record Dates: First submitted 2019-02-25; First posted 2019-03-05 (Actual); Last update posted 2019-03-05 (Actual); Status verified 2019-03

CONDITIONS: Chronic Periodontitis; Periodontal Bone Loss; Resistance Bacterial
Keywords: Periodontitis; Microbiome; Dysbiosis; Homeostasis; Dental plaque; Antibiotics
MeSH Terms: conditions — Chronic Periodontitis; Alveolar Bone Loss; Periodontitis; Dysbiosis; Dental Plaque | interventions — Weights and Measures; Root Planing

STUDY DESIGN:
Intervention Model Description: Double blinded, randomized clinical trial.
Who Masked: Participant, Care Provider
Masking Description: Double-blinding: The researchers who performed the measurements and treatment will be different from those who performed the microbial analysis; the examiner will be blinded during the entire duration of the study about the type of analysis subgingival dental plaque has been undergone.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- The exCELLigence system (Active Comparator): 1. Following the baseline examination each of the 20 randomly selected patients will be informed about the cause of periodontal disease.
  2. The 10 deepest interproximal sites in each quadrant will be selected and exposed to microbial sampling. Two sterilized paper points will be inserted into the pocket of each site and will be keep in place for 60 s. The twin paper points will be remove and distributed in two vials and transfer for microbiological processing.
  3. The study participants will undergo SCALE AND ROOT PLANING (SRP). SRP will be performed two quadrants at a time under local anaesthesia at approximately weekly intervals.
  4. The adjunctive antibiotics selected by 'the exCELLingence' system will be started at the second SRP visit.
  Interventions: Procedure: SCALE AND ROOT PLANING; Drug: ADJUNTIVE ANTIBIOTICS; Diagnostic Test: MICROBIAL SAMPLING
- Origen (Active Comparator): 1. Following the baseline examination each of the 20 randomly selected patients will be informed about the cause of periodontal disease.
  2. The 10 deepest interproximal sites in each quadrant will be selected and exposed to microbial sampling. Two sterilized paper points will be inserted into the pocket of each site and will be keep in place for 60 s. The twin paper points will be remove and distributed in two vials and transfer for microbiological processing.
  3. The study participants will undergo SCALE AND ROOT PLANING (SRP). SRP will be performed two quadrants at a time under local anaesthesia at approximately weekly intervals.
  4. The adjunctive antibiotics agents selected by 'Origen' laboratories analysis will be started at the second SRP visit.
  Interventions: Procedure: SCALE AND ROOT PLANING; Drug: ADJUNTIVE ANTIBIOTICS; Diagnostic Test: MICROBIAL SAMPLING
- Echevarne (Active Comparator): 1. Following the baseline examination each of the 20 randomly selected patients will be informed about the cause of periodontal disease.
  2. The 10 deepest interproximal sites in each quadrant will be selected and exposed to microbial sampling. Two sterilized paper points will be inserted into the pocket of each site and will be keep in place for 60 s. The twin paper points will be remove and distributed in two vials and transfer for microbiological processing.
  3. The study participants will undergo SCALE AND ROOT PLANING (SRP). SRP will be performed two quadrants at a time under local anaesthesia at approximately weekly intervals.
  4. The adjunctive antibiotics agents selected by 'Echevarne' laboratories analysis will be started at the second SRP visit.
  Interventions: Procedure: SCALE AND ROOT PLANING; Drug: ADJUNTIVE ANTIBIOTICS; Diagnostic Test: MICROBIAL SAMPLING

INTERVENTIONS:
Procedure: SCALE AND ROOT PLANING — SRP will be performed two quadrants at a time under local anaesthesia at approximately weekly intervals.
  Each session will be carried out with the following materials: - Ultrasound device (SONICflex 2003 / L) and curettes (Hu-Friedy Manufacturing, Illinois, USA).
Drug: ADJUNTIVE ANTIBIOTICS — The antimicrobial adjunctive agents selected by 'Echevarne' laboratories analysis will be started at the second SRP visit.
  The antibiotic will be selected among AMOXICILIN, METRONIDAZOLE, AMOXICILIN + METRONIDAZOLE AND AZITROMYCIN.
Diagnostic Test: MICROBIAL SAMPLING — 1. Before treatment, the 10 deepest interproximal sites in each quadrant will be selected and exposed to microbial sampling. Two sterilized paper points will be inserted into the pocket of each site and will be keep in place for 60 s. The twin paper points will be remove and distributed in two vials and transfer for microbiological processing.
  2. The subgingival microbiota will be harvested from the sampling sites 2 months after the completion of active therapy.

SUMMARY:
The aim of the study is to develop an in vitro model of growth of oral biofilms, and validate xCELLigence system for the selection of an effective antibiotic treatment for each patient.

DETAILED DESCRIPTION:
Periodontitis in a chronic disease caused by bacteria present in the subgingival flora, which induces an inflammatory response of periodontal tissues. It has been suggested that some periodontal pathogens may be inaccessible to mechanical periodontal therapy due to its ability to invade the gingival tissues and evade defense mechanisms of the host. Therefore, it is conceivable that coadjuvant administration of antimicrobials may improve the outcome of mechanical therapy. There are several techniques to monitor periodontal pathogens and determine antibiotic therapy. But the most important disadvantage of conventional laboratory methods is that they are indirect, based on the molecular detection of 3 to 10 bacterial species, without analyzing whether the biofilm as a whole is sensitive or resistant to treatment, being a possible cause of failure and / or recurrence of the disease, in addition to the risk of development of antimicrobial resistance.

The investigators hypothesis is that the specific selection of antimicrobial treatment with the xCELLigence system allows better improvements in clinical parameters than indirect laboratory methods.

Materials and methods:

A randomized double-blind clinical trial will be launched. Samples of subgingival plaque will be taken with paper tips. Subjects included in the study will be randomized to one of 3 treatment groups: scaling and root planing combined with systemically administration of antibiotic suggested by the xCELLigence system; scaling and root planing combined with systemically administration of antibiotic suggested by 'Echevarne' laboratory and scaling and root planing combined with systemically administration of antibiotic suggested by 'Origen' laboratory.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects of 40-70 years.
2. No smokers or smokers of less than 10 cigarettes a day.
3. Patients with periodontitis stages III and IV grades A-B.
4. Presence of 20 natural teeth, including at least three molar teeth.
5. Presence of at least 4 sites with at least 6 mm probing depth.
6. Good general health

Exclusion Criteria:

1. Smokers of more than 10 cigarettes a day.
2. Patients who have received periodontal treatment in the previous 12 months.
3. Patients who have used antibiotics in the last 6 months.
4. Routine use of oral antiseptics and / or during the previous 3 months.
5. Systemic conditions that required antibiotic premedication.
6. Women pregnant or nursing.
7. Medications that could influence the outcome of periodontal therapy.
8. Any known allergies to the test antimicrobial agents.
9. Diabetics.

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2019-02-08 (Actual); Primary Completion 2019-08 (Estimated); Study Completion 2019-08 (Estimated)

PRIMARY OUTCOMES:
Clinical measure: Clinical attachment loss (CAL) change | 1. Baseline, 2. Reevaluation (60 days after Scale and root planing).
  It is defined as the distance in millimeters between CEJ and the end of the periodontal pocket. The calculation of the depth of the pocket + gingival recession or pocket depth - gingival hyperplasia will be carried out.
Clinical measure: Probing pocket depth (PPD) change | 1. Baseline, 2. Reevaluation (60 days after Scale and root planing).
  The probing depth will be measured in six areas (disto-buccal, mediate-vestibular, mesio-buccal, disto-palatal, mid-palatal, and mesio-palatal) of each tooth with Williams PQ-OW 208 396 probe. It will be use with a pressure of 20 grams that is equivalent to the pressure of dropping the weight of the probe without exerting additional pressure.
Clinical measure: Bleeding on probing (BOP) change, Gingival Bleeding Index. | 1. Baseline, 2. Reevaluation (60 days after Scale and root planing).
  The "Full mouth bleeding score" (FMBS) will be calculated based on scores of 0 (no bleeding) or 1 (bleeding) after probing depths are checked. Four surfaces per tooth are evaluated: mesial, distal, vestibular and lingual.
O'leary plaque index change | 1. Baseline, 2. Reevaluation (60 days after Scale and root planing).
  The percentage of gingival surfaces with presence of plaque in the dentogingival junction of the teeth is found. Four surfaces per tooth are evaluated: mesial, distal, vestibular and lingual.

CONTACTS AND LOCATIONS:
Locations (1):
- Marta Reglero Santaolaya, Valencia, Spain